CLINICAL TRIAL: NCT02056600
Title: A Randomized, Open-label, Single Dose, Two-way Crossover Clinical Trial to Investigate the Pharmacokinetics and Safety/Tolerability of the Combination of Gemigliptin/Metformin HCl Sustained Release 50/1000mg in Comparison to Each Component Gemigliptin 50mg and Metformin HCl Extended Release 1000mg Administered in Healthy Male Volunteers
Brief Title: BE Study of the Combinations of Gemigliptin 50mg and Metformin HCl Extended Release 1000mg in Comparison to Each Component Administered Alone.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LG Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: LG-DMCL004
Record Dates: First submitted 2014-02-05; First posted 2014-02-06 (Estimated); Last update posted 2014-05-08 (Estimated); Status verified 2014-05

CONDITIONS: Healthy
MeSH Terms: interventions — LC15-0444

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- G+M (Experimental): Coadministration of gemigliptin 50mg and metformin HCl extended release 1000mg
  Interventions: Drug: gemigliptin and metformin HCl extended release
- C (Experimental): Combination of gemigliptin50mg/metformin HCl sustained release 1000mg
  Interventions: Drug: gemigliptin/metformin HCl sustained release

INTERVENTIONS:
Drug: gemigliptin and metformin HCl extended release — Coadministration of gemigliptin 50mg and metformin HCl extended release 1000mg, for 1 day
  Arms: G+M
Drug: gemigliptin/metformin HCl sustained release — Administration of combination of gemigliptin 50mg/metformin HCl sustained release 1000mg, for 1day.
  Arms: C

SUMMARY:
This study is to evaluate the safety/tolerability and pharmacokinetics of the combinations of gemigliptin 50mg and metformin HCl extended release 1000mg in comparison to each component administered in healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male adults at age between 20 to 45 at the time of the screening
* ThoseSubjects whose BMI measurement at screening visit is between 18 and 27 kg/m2
* Subjects with fasting plasma glucose (FPG) of 70-125 mg/dL at screening visit
* Subject who has voluntarily decided to participate in this clinical trial and onsented in writing

Exclusion Criteria:

* Subjects who have a past or present clinically significant disease such as hepatic, renal, gastrointestinal, respiratory, musculoskeletal, endocrine, neurological, hemato-oncological, or cardiovascular disorder
* Subjects who have a past history of gastrointestinal disease (e.g. Crohn's disease, ulcer, etc.) or surgery (however, simple appendectomy and hernioplasty are not included) that can affect the absorption of drugs
* Subjects with a medical history of allergic reaction to other drugs including the investigational products or clinically significant hypersensitivity reaction
* Subjects who have a history of drug abuse
* Subjects who have shown positive reaction to drugs that may be abused from a urine drug screening
* Subjects who took other investigational product in other trials within 90 days before the first administration of this investigational product
* Subjects who had whole blood donation within 60 days or component blood donation within 30 days before the first administration of the investigational product, or transfusion within 30 days before the first administration
* Subjects who have taken a drug which is expected to have an effect on the clinical trial within 14 days before the date of the first administration of the investigational product or have had any food that is expected to have an effect on the clinical trial within 7 days (e.g. drinks containing caffeine, grapefruit juice, etc.)
* Subjects who have had alcohol containing drinks 3 times or more per week within one month before the screening visit or cannot abstain from drinking after completing the informed consent form for the participation in the study to the end of the clinical trial
* Subjects who have smoker more than 10 cigarettes per day within the recent one month at the screening visit or cannot refrain from smoking the clinical trial period
* In the vital signs measured in sitting position at the screening visit, subjects who have showed a systolic blood pressure of < 90 mmHg or > 145 mmHg, a diastolic blood pressure of > 95 mmHg or < 60 mmHg) , or a pulse rate of > 110 bpm or < 40 bpm
* Subjects who showed the following findings in the tests conducted during the screening period:
* In excess of 1.5 times the upper normal limit (UNL) in hepatic enzyme (AST and ALT) values
* The creatinine clearance calculated by Cockcroft-Gault equation is 80 mL/min or less
* Positive result in serum test (hepatitis type B test, hepatitis type C test, Human Immunodeficiency Virus (HIV) test, syphilis test)
* QTc > 450 msec in ECG or a clinically significant abnormal rhythm
* Subjects who are considered to be unsuitable in conducting the clinical trial for other reason at the principal investigator's discretionary judgment

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2014-03; Primary Completion 2014-04 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
AUClast | up to 48h post-dose
  To evaluate AUClast of gemigliptin and metformin
Cmax | up to 48h post-dose
  To evaluate Cmax of gemigliptin and metformin

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Cho YS, Lee SH, Lim HS, Bae KS. Pharmacokinetic Equivalence of the High Dose Strength Fixed-Dose Combination Tablet of Gemigliptin/Metformin Sustained Release (SR) and Individual Component Gemigliptin and Metformin XR Tablets in Healthy Subjects. J Korean Med Sci. 2018 Sep 5;33(41):e258. doi: 10.3346/jkms.2018.33.e258. eCollection 2018 Oct 8. PMID 30288156